CLINICAL TRIAL: NCT05599971
Title: The Efficacy of Intralesional Injection of Combined Digoxin and Furosemide Versus 5-Flurouracil in the Treatment of Plantar Warts
Brief Title: Intralesional Injection of Combined Digoxin and Furosemide Versus 5-Flurouracil in Plantar Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Norhan Anees, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: planter wart treatment
Record Dates: First submitted 2022-10-19; First posted 2022-10-31 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Plantar Wart
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): 15 patients will receive intralesional 0.1 mL of combined digoxin and furosemide, with maximum 5 warts per session.
  Interventions: Drug: intralesional combined digoxin and furosemide
- Group B (Active Comparator): 15 patients will receive intralesional injection of 5- Fluorouracil (50mg/ml) in full concentration into the wart using a 27- gauge insulin syringe till the entire lesion begins to puff up. The maximum dose injected per session will be 2ml of 5-FU.
  Interventions: Drug: intralesional injection of 5- Fluorouracil
- Group c (Placebo Comparator): 15 patients will receive intralesional saline.
  Interventions: Other: intralesional saline

INTERVENTIONS:
Drug: intralesional combined digoxin and furosemide — 15 patients will receive intralesional combined digoxin and furosemide, with maximum 5 warts per session. 0.2 mL of lignocaine (20 mg/mL) will be used as a local analgesic and after few minutes, 0.1 mL of combined digoxin and furosemide solution will be slowly injected into the base of each wart. Selected patients will receive one session every 2 weeks till complete clearance or up to 5 sessions.
  Arms: Group A
Drug: intralesional injection of 5- Fluorouracil — 15 patients will receive intralesional injection of 5- Fluorouracil (50mg/ml) in full concentration into the wart using a 27- gauge insulin syringe till the entire lesion begins to puff up. The maximum dose injected per session will be 2ml of 5-FU. Selected patients will receive one session every 2 weeks till complete clearance or up to 5 sessions.
  Arms: Group B
Other: intralesional saline — 15 patients will receive intralesional saline. Selected patients will receive one session every 2 weeks till complete clearance or up to 5 sessions.
  Arms: Group c

SUMMARY:
The aim of the current work is to evaluate the efficacy and safety of intralesional combined Digoxin and furosemide versus intralesional 5-flurouracil in the treatment of plantar warts.

DETAILED DESCRIPTION:
Warts are benign proliferations of skin and mucosa caused by the human papilloma virus (HPV). Currently, over 170 HPV types have been identified. Certain HPV types tend to infect skin at specific anatomical sites, such as palmoplantar warts, which are typically caused by serotypes 1, 2, and 4, however warts caused by any HPV type can occur at any site (Tulay & Serakinci, 2016).

Plantar warts most commonly present with pain that occur with activities that put pressure on the soles of the feet. They commonly affect plantar areas of increased pressure, such as the heels or metatarsal heads. On gross inspection, plantar warts may appear as a singular rough, flesh-colored to yellow or grey-brown, hyperkeratotic papule, or a thickened "cobblestoned" plaque, termed a mosaic wart, which consists of multiple plantar warts that have coalesced (Witchey et al., 2018).

There are several modalities for the treatment of warts including, cryotherapy, electrocoagulation, topical salicylic acid, topical 5-fluorouracil, intralesional immunotherapy, and laser surgery. All these treatment options can be painful, time-consuming, and/or expensive, and none is considered the gold standard (Latif et al., 2021).

K+ influx is essential for the replication of DNA viruses, such as HPV. Both digoxin, which is a cardiac glycoside, and furosemide, which is a loop diuretic, inhibit the K+ influx by interacting with cell membrane ion co-transporters (Na+/K+-ATPase and Na+-K+-2Cl-co-transporter-1). Therefore, it is hypothesized that these two compounds may be valuable in the treatment of HPV-induced warts. This new approach is called ionic contra-viral therapy (Rijsbergen et al., 2019). Intralesional injection of combined digoxin and furosemide was found to be safe and effective as a treatment option for multiple plantar warts (Fathy et al., 2021).

5-Fluorouracil (5-FU) is an antimetabolite that can be used alone or with other chemotherapeutic agents to treat solid tumors. It is one of the pyrimidine analogues. Due to its structure, 5-FU disrupts nucleoside metabolism and can be integrated into the single and double helix of RNA and DNA, respectively, causing cell cytotoxicity and death (Zoheir et al., 2022).

Intralesional 5-fluorouarcil has been found to be a highly effective, safe and cheap alternative in the treatment of warts, with a significantly good response in genital warts also (Kamal et al., 2108).

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple plantar warts (≥ 3) will be included.

Exclusion Criteria:

* Patients under 18 years old or patients over 65 years old.
* Pregnancy or breast feeding.
* Patients received vaccination or any other treatment of warts during the last month.
* Patients with a known sensitivity to any of the investigational product ingredients.
* Patients with history of asthma, allergic skin disorders or convulsions.
* Patients with signs of any systemic or local inflammation or infection.
* Patients with any evidence of immunosuppression including HIV.
* History of cardiac diseases, relevant abnormal K level or ECG abnormalities for patients who will receive the combined digoxin and furosemide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-22 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
change in size of the warts | through study completion, an average of 9 months
  The studied warts will be clinically evaluated regarding change in size
Dermoscopic evaluation | through study completion, an average of 9 months
  The patients will be categorized in to 4 scores according to their response to treatment as:
  Score 0: patients showed neither clinical response nor dermoscopic clearance of warts 2 weeks after the last treatment session.
  Score 1: patients showed clinical improvement with decreased size of wart and thickness of callus without dermoscopic clearance of warts 2 weeks after the last treatment session.
  Score 2: patients showed disappearance of warts clinically (clinical clearance) but dermoscopic examination revealed remnants of warts 2 weeks after the last treatment session.
  Score 3: patients showed clinical and dermoscopic clearance of warts 2 weeks after the last treatment session (Barkat et al., 2018).
treatment-related adverse effects | through study completion, an average of 9 months
  Immediate and late adverse effects will be evaluated
Patients' satisfaction | through study completion, an average of 9 months
  Patients' satisfaction will be evaluated through a questionnaire. Patients' satisfaction will be graded into (very satisfied, satisfied, and unsatisfied).

REFERENCES:
- See also: Related Info — https://scholar.google.com.eg/scholar?hl=ar&as_sdt=0%2C5&q=https%3A%2F%2Fonlinelibrary.wiley.com%2Fdoi%2Ffull%2F10.1111%2Fijd.14092&btnG=
- See also: Related Info — https://scholar.google.com.eg/scholar?hl=ar&as_sdt=0%2C5&q=https%3A%2F%2Fonlinelibrary.wiley.com%2Fdoi%2Ffull%2F10.1111%2Fjocd.13913&btnG=
- See also: Related Info — http://www.jpad.com.pk/index.php/jpad/article/view/1267
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8906267/
- See also: Related Info — https://scholar.google.com.eg/scholar?hl=ar&as_sdt=0%2C5&q=https%3A%2F%2Fonlinelibrary.wiley.com%2Fdoi%2Ffull%2F10.1111%2Fbjd.17583&btnG=
- See also: Related Info — https://jcmtjournal.com/article/view/1533
- See also: Related Info — https://www.degruyter.com/document/doi/10.7556/jaoa.2018.024/html
- See also: Related Info — https://scholar.google.com.eg/scholar?hl=ar&as_sdt=0%2C5&q=https%3A%2F%2Faimj.journals.ekb.eg%2Farticle_231304.html&btnG=